CLINICAL TRIAL: NCT04792528
Title: Repeated Advanced Cognitive Training in Mild Cognitive Impairment (The REACT MCI Study). A Randomized, Controlled Trial.
Brief Title: REACT MCI - Repeated Advanced Cognitive Training in Mild Cognitive Impairment
Acronym: REACT MCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Oslo University Hospital (Other); NKS Olaviken (Unknown); St. Olavs Hospital (Other); NKS Kloverasen (Unknown); Barrow Neurological Institute (Other); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 77084 REACT MCI; Prosjektnr. 2019208 (Other Grant/Funding Number: Program for klinisk forskningsbehandling (KLINBEFORSK))
Record Dates: First submitted 2021-02-23; First posted 2021-03-11 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment
Keywords: computer-based cognitive training
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomization in blocks of six to eight will be performed by the regional research support statistics service to either two training periods, one training period or generalized brain training/active control.
Who Masked: Investigator
Masking Description: All study personnel except for the PI, coaches and Study secretary will be blinded for group allocation regarding types of memory training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One training period (Experimental): One training period of 30 minutes of daily adaptive training for 4-5 days a week up for 20- 25 trainings using computerized cognitive training.
  Interventions: Other: Computerized cognitive training.
- Two training periods (Experimental): Two training periods of 30 minutes of daily adaptive training for 4-5 days a week up for 20- 25 trainings using computerized cognitive training.
  Interventions: Other: Computerized cognitive training.
- Active control (Active Comparator): The generalized brain training group (Active control) will play solitaire 30 minutes daily for 25 sessions
  Interventions: Other: Generalized brain training / Active control

INTERVENTIONS:
Other: Computerized cognitive training. — COGMED RM program (Pearson Inc., UK)
  Arms: One training period; Two training periods
Other: Generalized brain training / Active control — Solitaire
  Arms: Active control

SUMMARY:
Background:

Dementia is a debilitating and devastating disease impacting the individuals, their families, and the health care system. According to the World Health Organization the dementia epidemic could overwhelm the global health care system and undermine social and economic development. Currently, no curative treatment for dementia exists despite immense research activity.

The cognitive and functional impairment in dementia, especially Alzheimer's disease (AD), develop slowly decades before clinical signs emerge. This knowledge has led to the recognition of a prodromal period of mild cognitive impairment (MCI), between normal cognition and dementia. This is at present the earliest stage for intervention in dementia; even a short delay in dementia progression will have a large impact on global economy and health care.

Objectives:

In this clinical multicenter study, we aim to investigate the efficiency and cost-effectiveness of working memory training in MCI. To identify high responders to training analysis of genetic markers, relative's stress and craniospinal clearance will be performed.

Participants and methods:

This study is a blinded, randomized and controlled trail that will include 213 participants, diagnosed with MCI, included from five Norwegian Memory clinics in four health care regions. The groups will be randomized to either two training periods, one training period or active control. The intervention is computerized working memory training. Neuropsychological status, activities of daily living (ADL), and relative stress and quality of life will be assessed at baseline and 3, 6, 12 ,24 and 48 months after training. Structural MRI will be performed at baseline, and 3 and 6 months after training.

For participants in the REACT MCI glymphatics substudy craniospinal clearance will be measured at baseline.

A cost-utility analysis will be performed to evaluate if the working memory training is more cost-effective compared to the active control group in the MCI phase, taking a societal perspective.

ELIGIBILITY:
Inclusion Criteria for the REACT MCI study:

* Diagnosis of MCI, based on the Mayo/winblad criteria or confirmation of current MCI status within the last 6 months before study enrollment.
* The ability to use and accessibility to an iPad or computer.
* Fluent in Norwegian.
* Spinal tap performed and results available

Exclusion Criteria for the REACT MCI study:

* Patients unable to undergo a MRI investigation based on claustrophobia or metal foreign bodies are excluded from the study.
* Major psychiatric illness and current substance abuse
* Recent stroke

Inclusion Criteria for the REACT MCI Glymphatics substudy:

* Enrollment in the REACT MCI study
* Participant allocated to Sorlandet Hospital or Oslo University Hospital

Exclusion Criteria for the REACT MCI Glymphatics substudy:

* Individuals with known allergy against contrast solutions
* Individuals with other serious allergies
* Individuals with kidney failure or glomerular filtration rate < 30
* Individuals younger than 18 or older than 80
* Pregnant or lactating women
* For individuals >70 years or with medications affecting kidney function the glomerular filtration rate needs to be less than week old.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2028-10-25 (Estimated)

PRIMARY OUTCOMES:
Working memory training is superior to active control measured by spatial span backwards at 6 months | From enrollment until 6 months
Reduced function in the glymphatic system is associated with reduced working memory training effect measured by CT evaluated craniospinal clearance | Enrollment to 12 months
  Craniospinal clearance will be evaluated with a single CT image scan at level with the foramen magnum.
Working memory training impact quality of life measure in the participants as compared to active control measured by EuroQOL5D-5L after 12 months. | Enrollment to12 months
Working memory training prolongs the MCI phase as compared to active controls | Enrollment to 48 months
  We consider the participants as having dementia when they no longer rapport intact activities of daily living and in addition display reduction of 1.5 standard deviation on test score on two tests on three or more cognitive domains.

SECONDARY OUTCOMES:
The effect of working memory training is dose related measured by spatial span backwards after 6 months | Enrollment to 6 months
Allelic variations in predefined genetic markes influence training effects after 3 months measured by spatial span backwards. | Enrollment to 3 months
  Allelic variations of LMX1a, APOE, AQP4 and/or COMT have in previous publications shown variable impact on working memory training. A statistical model combining these genes will be fitted for this investigation
Workin memory training reduces relatives stress scores as compared to relatives stress scores in the active control group after 12 months | Enrollment to 12 months
  Relatives stress score (RSS) is a validated scale measuring the stress for relatives
Working memory training reduces QALY associated cost as compared to active controls at 24 months. | Enrollment to 24 months
  The generic outcome in the analysis is QALYs (Quality adjusted life years) derived from the instrument EQ-5D 5L. The second outcome is production loss of the relatives and patients associated with MCI through the progression of dementia The health economic analysis will include following costs: 1) intervention related costs 2) direct costs/health care costs, mainly related to use of health care services, including primary, secondary and tertiary care and health services 3) indirect costs, including work absence for the patients and the relatives of the patients (i.e., productivity loss). Data will be collected through a self-report measures (EQ-5D 5L), and from the Norwegian patient registry.
Working memory training reduces QALY associated cost as compared to active controls at 48 months. | enrollment to 48 months
  The generic outcome in the analysis is QALYs (Quality adjusted life years) derived from the instrument EQ-5D 5L. The second outcome is production loss of the relatives and patients associated with MCI through the progression of dementia The health economic analysis will include following costs: 1) intervention related costs 2) direct costs/health care costs, mainly related to use of health care services, including primary, secondary and tertiary care and health services 3) indirect costs, including work absence for the patients and the relatives of the patients (i.e., productivity loss). Data will be collected through a self-report measures (EQ-5D 5L), and from the Norwegian patient registry.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne S Hernes, M.D. Phd., Principal Investigator — Sørlandet Sykehus HF, Universitetet i Bergen
Locations (5):
- Norway (5):
  - Sørlandet Sykehus Arendal, Arendal
  - NKS Olaviken Alderspsykiatriske sykehus - Hukommelsesklinikk, Bergen
  - N.K.S. Kløveråsen, Bodø
  - Oslo Universitetssykehus Ullevål, Oslo
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No